CLINICAL TRIAL: NCT04730323
Title: TOCILIZUMAB - An Option for Patients With COVID-19 Associated Cytokine Release Syndrome; A Single Center Experience
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FMH College of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Aijaz Zeeshan Khan Chachar, Consultant Physician (Senior Registrar), FMH College of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# FMH-05-2020-IRB-75
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Tocilizumab; Covid-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tocilizumab Group (Experimental): Tocilizumab administration protocol: Patients received an initial dose calculated as per the body weight (8mg/kg) maximum 800mg/dose) over 1 hour, followed by up to three additional doses if required as per the response after the first dose with 8 hours intervals. Predefined Parameters of disease severity were assessed 12 to 24 hourly. Injection Paracetamol 1g was administered before infusion.
  Interventions: Drug: Tocilizumab
- Methylprednisolone (corticosteroid) group (Active Comparator): Corticosteroid administration protocol: Patients received methylprednisolone 80mg/day in two divided doses as per national/local guidelines and predefined parameters of disease severity were assessed on each day.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants received an initial dose calculated as per the body weight (8mg/kg) maximum 800mg/dose) over 1 hour, followed by up to three additional doses if required as per the response after the first dose with 8 hours intervals. Predefined Parameters of disease severity were assessed 12 to 24 hourly. Injection Paracetamol 1g was administered before infusion. The response of the participants after Tocilizumab administration was recorded based on clinical parameters (Oxygen requirement, Fever, Need for invasive positive pressure ventilation), biochemical parameters (D-dimers, C-reactive protein (CRP), Ferritin, Lactate dehydrogenase (LDH) levels), Chest X-ray findings, and Repeated PCR test for COVID-19. Any side effects noted after administration of TOCILIZUMAB were recorded.
  Any side effects noted after administration of TCZ/ Corticosteroid were recorded.
  Other Names: Experimental

SUMMARY:
Investigators conducted this study to see the effectiveness of Tocilizumab in COVID-19 participants who were in cytokine release syndrome and there was also a control group who received steroids(RECOVERY TRIAL wasn't published or available at that time) this study was conducted in the early days of 1st wave of COVID in our country Pakistan so it was need of the day to develop some national guidelines on the basis of multiple studies' results from Pakistan.

DETAILED DESCRIPTION:
Objectives: To analyze the effectiveness of Tocilizumab in moderate to severe Covid-19 participants on the basis of predefined assessment criteria.

Study Settings: Single center, Fatima Memorial Hospital, Lahore.

Study Design: Quasi experimental.

Duration of Study: From 12th May, 2020 to 12th July, 2020.

Participants & Methods: Sample size and technique: Sample size was 93; 33 participants were kept in experimental group, given Tocilizumab, 8mg/kg intravenously or 162 mg subcutaneously and rest of the 60 participants were given corticosteroids, methylprednisolone 80 mg/day. Consecutive sampling.

Failure of therapy was labeled when participants were intubated or died, and the endpoints were failure-free survival which was the primary endpoint and overall survival secondary at the time of discharge.

ELIGIBILITY:
* Inclusion Criteria:

  * All patients diagnosed with COVID-19 infection with positive reverse transcriptase RT-PCR test, willing to participate in this study or PCR negative patients with clinically COVID-19 Pneumonia in cytokine storm as evidenced by raised inflammatory markers with typical radiological changes
  * Patients of both genders were included
  * Patients having an age of > 65 years with proven Cardiomyopathy, Coronary artery disease, chronic lung disease, Immunosuppressed or organ transplant End-stage renal disease on history & examination and medical records and having any 1 out of 4 Fever 0f
  * ≥39 C
  * Hypotension or drop in mean arterial pressure of > 10mmHg
  * Progressive Hypoxemia requiring > 5 liters of oxygen
  * Sustained Respiratory rate >30/min with any 2 laboratory parameters out of 3 are present D-dimers ≥ 1000 ng/ml C-reactive protein CRP ≥ 100mg/L Ferritin ≥ 600ng/ml
  * Patients having low risk or no comorbidities and having an age of <65 years with having any 3 out of 4 Fever 0f
  * ≥39 C
  * Hypotension or drop in mean arterial pressure of > 10mmHg
  * Progressive Hypoxemia requiring > 5 liters of oxygen
  * Sustained Respiratory rate >30/min With any 2 laboratory parameters out of 3 are present D-dimers ≥ 1000 ng/ml C-reactive protein CRP ≥ 100mg/L Ferritin ≥ 600ng/ml
  * Moderate severe or severe COVID 19 features

    1. Shortness of breath oxygen saturation <93% on room air
    2. Progressive Hypoxemia requiring > 5 liters of oxygen
    3. Respiratory rate >30/min
    4. The partial pressure of arterial oxygen to fraction of inspired oxygen ratio<300
    5. Lung infiltrates on Chest x-ray CXR >50% within 24 to 48 hrs
    6. Respiratory failure
* Exclusion Criteria:

  * Known severe allergic reactions to Tocilizumab or any other monoclonal antibody
  * Pregnancy or breastfeeding
  * Absolute Neutrophil Count(ANC) < 1000
  * Alanine aminotransferase(ALT) or aspartate aminotransferase (AST) > 5 times upper normal limit
  * Platelet count of < 50,000
  * Bowel diverticulitis or bowel perforation
  * Patients having Acute pancreatitis

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Decreased Mortality in Participants | 30 days
  investigators tried to find out that whether there is decreased mortality in expermiental and active Comparator group or not
Hospital & ICU stay in days | 14 days
  investigators tried to find out that whether there is decreased hospital and ICU stay in experimental group & active Comparator

CONTACTS AND LOCATIONS:
Overall Officials: Aijaz Zeeshan Khan Chachar, MBBS,FCPS, Study Director — FMH College of Medicine & Dentistry
Locations (1):
- Fatima Memorial Hospital College of Medicine & Dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared with researchers in future too
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Whenever will be asked to, within few days
Access Criteria: Only officials can access the data

REFERENCES:
- [Derived] Chachar AZK, Khan KA, Iqbal J, Shahid AH, Asif M, Fatima SA, Khan AA, Younis BB. "Tocilizumab-an option for patients with COVID-19 associated cytokine release syndrome: A single center experience", a retrospective study-original article. Ann Med Surg (Lond). 2021 Mar;63:102165. doi: 10.1016/j.amsu.2021.02.011. Epub 2021 Feb 8. PMID 33585031

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT04730323/Prot_SAP_000.pdf